CLINICAL TRIAL: NCT02273713
Title: The ACTION Trial: a Phase Ib/II Study on the Addition of Nab-paclitaxel (Abraxane) to Capecitabine and Oxaliplatin in the First-line Treatment of Metastasized Oesophagogastric Carcinoma.
Brief Title: The Addition of Nab-paclitaxel (Abraxane) to First Line Treatment of Metastasized Oesophagogastric Carcinoma (ACTION)
Acronym: ACTION
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL 49837.018.14
Record Dates: First submitted 2014-10-17; First posted 2014-10-24 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Cancer; Toxicity
Keywords: Esophageal cancer; Metastasized; Nab-paclitaxel; Toxicity; First line treatment; Phase Ib/II
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-Paclitaxel (Experimental): Nab-Paclitaxel added to first line treatment with Oxaliplatin and Capecitabine
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel added to first line treatment oxaliplatin and capecitabine
  Other Names: Abraxane

SUMMARY:
Oesophagogastric cancer is a major cause of cancer related mortality, with an overall 5-year survival rate of 10% worldwide and patients are often diagnosed with locally advanced or metastasized disease at first presentation. For advanced oesophagogastric cancer fluoropyrimidines are the backbone of palliative chemotherapy and is commonly used in 2- or 3-drug combinations .

However, in clinical practice after progression on first line therapy, a substantial number of oesophagogastric cancer patients may not be able to start second line chemotherapy due to rapid clinical deterioration. Therefore, new triplets with high anti-tumor activity and low toxicity are urgently needed.

Given the activity of capecitabine and oxaliplatin containing regimens and the potential of taxanes in oesophagogastric cancer, the investigators propose a phase I study combining capecitabine and oxaliplatin with Nab-paclitaxel.

Solvent-based taxanes (paclitaxel, docetaxel) can cause severe toxicities not only by the active agents itself but also by the solvents like cremophor. Nab-paclitaxel (Abraxane) is a solvent-free formulation of paclitaxel encapsulated in albumin. It does not require premedication with corticosteroids or antihistamines to prevent the risk of solvent-mediated hypersensitivity reactions. This new formulation improves safety profile, allows higher dosing with shorter infusion duration, and produces higher tumor drug concentration. It has proven activity in breast cancer, non small lung cancer and pancreatic cancer, as well as in gastric cancer models.

DETAILED DESCRIPTION:
Phase 1: To assess the safety and tolerability of Nab-paclitaxel added to oxaliplatin and capecitabine at their currently optimal doses.

Phase 2: To determine the anti-tumor activity of Nab-paclitaxel when co-administered with oxaliplatin and capecitabine in patients with irresectable or metastasized oesophagogastric cancer in terms of progression free survival.

Study design This is a single-center, open label, dose finding, phase I/II study.

Intervention In the phase I part of the study, the dose of nab-paclitaxel in combination of capecitabine and oxaliplatin will be escalated in fixed increments according to the dose escalation scheme outlined below

Dose level Nab-paclitaxel Capecitabine Oxaliplatin Minimum Day 1 and 8 14 days Day 1 and 8 number of patients -1 40 mg/m2 1000 mg/m2 65 mg/m2 -

1. (starting) 60 mg/m2 1000 mg/m2 65 mg/m2 3
2. 80 mg/ m2 1000 mg/m2 65 mg/m2 3
3. 100 mg/ m2 1000 mg/m2 65 mg/m2 3
4. 120 mg/ m2 1000 mg/m2 65 mg/m2 3

In the phase II part of the study the maximum tolerated dose from the phase I part of the study will be used in combination with fixed dosages of capecitabine and oxaliplatin; nab-paclitaxel day 1 and 8 according to the Maximum Tolerated Dose (MTD) of the phase 1 part of the study combined with capecitabine for 14 days at 1000mg/m2 twice daily and oxaliplatin day 1 and 8 65mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent according to ICH/GCP, and national/local regulations prior to any screening procedures.
* Patients with histologically confirmed diagnosis of metastatic or irresectable carcinoma of the stomach or oesophagus
* Patients with metastatic or irresectable carcinoma of the stomach or oesophagus not pre-treated with chemotherapy or radiotherapy for irresectable or metastatic disease.
* Measurable disease as assessed by RECIST 1.1
* ECOG (WHO) performance status 0-2
* Patient has adequate bone marrow and organ function
* If a female patient is of child-bearing potential: negative serum pregnancy test, If sexually active, the patient must agree to use contraception.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Prior systemic treatment for metastatic or irresectable stomach or oesophageal cancer.
* Evidence of disease progression within 3 months after completion of adjuvant or neoadjuvant treatment containing capecitabine and/or oxaliplatin.
* History of hypersensitivity to nab-paclitaxel, capecitabine or oxaliplatin.
* All target lesions in a radiation field without documented disease progression.
* WHO 2-4
* Use of other investigational drugs within 30 days of enrollment.
* Patient has known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no oedema, no steroids and stable in 2 scans at least 4 weeks apart).
* History of malignancy in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
* Patients who are not willing to avoid consumption of Seville oranges, grapefruit or grapefruit juice grapefruit hybrids, pomelos and exotic citrus fruits during the entire study.
* Patient is currently being treated with drugs known to be strong inhibitors or inducers of CYP3A4 or CYP2C8, which cannot be discontinued or switched to a different medication 7 days prior to starting study treatment and for the duration of the study.
* Patient has active, uncontrolled bacterial, viral or fungal infection(s) requiring systemic therapy.
* Patient has known historical or active infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate patient participation in the clinical study (e.g. hematological, cardiovascular, lung disease etc)
* Patient is enrolled in any other clinical protocol or investigational trial with the same primary endpoint.
* Patients who in the investigators' opinion may be unwilling, unable or unlikely to comply with requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 12 months
  Identifying the Maximum Tolerated Dose
Progression Free survival | approximately 36 months

SECONDARY OUTCOMES:
Adverse events | approximately 36 months
  Adverse event, serious adverse events according to NCI CTC version 4.0
Response rate | approximately 36 months
  Response rate according to RECIST 1.1
Progression free survival | approximately 36 months
Neurotoxicity | approximately 36 months
  Self reported neurotoxicity according to EORTC QLQ CIPN20
Overall survival | approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, Prof.Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Medical Oncology, Amsterdam, Netherlands